CLINICAL TRIAL: NCT00459836
Title: A Phase Ib, Multi-Center, Open-Label, Dose Escalation Trial of Intravenous PR-104 Given in Combination With Docetaxel or Gemcitabine in Subjects With Solid Tumors
Brief Title: PR-104 and Docetaxel or Gemcitabine in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Brenda Gibson, Assoc. Director, Proacta, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-1003; PROACTA-PR-104-1003; PROACTA-WIRB-20070094
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — PR-104; Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: PR-104
Drug: docetaxel
Drug: gemcitabine hydrochloride
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as PR-104, docetaxel, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of PR-104 when given together with docetaxel or gemcitabine in treating patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of PR-104 in combination with docetaxel or gemcitabine hydrochloride in patients with solid tumors.

Secondary

* Determine the safety of PR-104 in combination with docetaxel or gemcitabine hydrochloride in these patients.
* Determine the antitumor activity of these regimens using disease-specific parameters, such as exams, scans, and tumor markers, in these patients.
* Determine the pharmacokinetics of PR-104 and its alcohol metabolite in these patients.
* Determine the pharmacokinetics of docetaxel and gemcitabine hydrochloride when administered with PR-104.
* Collect plasma samples for assessment of potential biomarkers of tumor hypoxia from these patients.
* Examine metabolic changes in tumors using fludeoxyglucose F 18 positron emission tomography (PET) and PET imaging with fluoromisonidazole F 18 (a hypoxia-targeted radiopharmaceutical) in these patients.

OUTLINE: This is a nonrandomized, open-label, uncontrolled, multicenter, dose-escalation study of PR-104. Patients are assigned to 1 of 2 treatment groups according to patient's malignancy and prior treatment history.

* Group 1: Patients receive docetaxel IV over 60 minutes and PR-104 IV over 60 minutes on day 1.
* Group 2: Patients receive gemcitabine hydrochloride IV over 30 minutes and PR-104 IV over 60 minutes on days 1 and 8.

In both groups, treatment repeats every 21 days for up to 8 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients in each group receive escalating doses of PR-104 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Blood is collected at baseline and periodically during course 1 for pharmacokinetic analysis. Plasma samples are analyzed for biomarkers of tumor hypoxia at baseline and on days 2 and 8.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor malignancy
* Treatment with either docetaxel or gemcitabine hydrochloride in combination with an investigational agent is reasonable
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL (red blood cell transfusion allowed)
* Bilirubin normal
* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* PT/INR or aPTT ≤ 1.1 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study therapy
* No evidence of any other significant medical disorder, including uncontrolled infection or infection requiring a concurrent parenteral antibiotic, or laboratory finding that, in the opinion of the investigator, would preclude study compliance
* No known HIV positivity
* No hepatitis B surface antigen positivity
* No hepatitis C positivity with abnormal liver function test

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to > 25% of bone marrow
* No prior high-dose chemotherapy (including conditioning for either myeloablative or nonmyeloablative transplantation)
* No more than 3 prior chemotherapy regimens
* More than 4 weeks since prior major surgery
* More than 4 weeks since prior investigational or traditional anticancer therapy (including radiotherapy) (6 weeks for nitrosoureas and mitomycin C)
* The following medications/treatments are not permitted during the trial:

  * Any other licensed or investigational anticancer treatment
  * Prophylactic hematopoietic growth factors
  * Irradiation therapy (palliative or therapeutic) unless given in the absence of tumor progression
* Concurrent systemic steroids allowed provided the patient is on a stable dose for ≥ 2 weeks prior to study treatment
* Concurrent androgen-deprivation therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-02; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of PR-104

SECONDARY OUTCOMES:
Safety of PR-104 as measured by CTCAE v3.0 criteria
Dose-limiting toxicity of PR-104
Pharmacokinetics of PR-104 and its alcohol metabolite in the blood
Pharmacokinetics of gemcitabine and docetaxel in the presence of PR-104
Antitumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Terri J. Melink, NP, MSN, ANP, Study Chair — Proacta, Incorporated
Locations (3):
- Proacta, Incorporated, San Diego, California, United States
- New Zealand (2):
  - University of Auckland Cancer Center, Auckland
  - Waikato Hospital, Hamilton

REFERENCES:
- [Derived] McKeage MJ, Jameson MB, Ramanathan RK, Rajendran J, Gu Y, Wilson WR, Melink TJ, Tchekmedyian NS. PR-104 a bioreductive pre-prodrug combined with gemcitabine or docetaxel in a phase Ib study of patients with advanced solid tumours. BMC Cancer. 2012 Oct 25;12:496. doi: 10.1186/1471-2407-12-496. PMID 23098625